CLINICAL TRIAL: NCT00019500
Title: A Randomized Phase II Trial of Two Doses of Raloxifene in Pre-Menopausal Women at High Risk For Developing Invasive Breast Cancer
Brief Title: Raloxifene in Preventing Breast Cancer in Premenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Prevention
Other Study IDs: CDR0000066428; NCI-98-C-0123; MB-402; NCT00001700 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2005-06-23 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2009-04

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Raloxifene Hydrochloride

INTERVENTIONS:
Drug: raloxifene
Procedure: evaluation of cancer risk factors

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of raloxifene may be an effective way to prevent breast cancer in premenopausal women.

PURPOSE: Phase II trial to study the effectiveness of raloxifene in preventing invasive breast cancer in premenopausal women.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of raloxifene in premenopausal women at high risk of developing invasive breast cancer.
* Determine the effect of raloxifene on blood steroid hormone levels (luteinizing hormone, estradiol, progesterone) and carotenoid levels during the menstrual cycle in these participants.
* Determine the effect of raloxifene on the endometrium and ovaries in these participants.
* Determine the effect of raloxifene on biochemical markers of bone metabolism, lipid profiles, and fibrinogen in these participants.
* Determine the effect of raloxifene on health-related quality of life of these participants.
* Determine the effect of raloxifene on bone mineral density in the spine and hip of these participants.

OUTLINE: This is an open-label study.

Participants are medically evaluated, followed by an observation period of 1 to 2 menstrual cycles. After the observation period, participants receive oral raloxifene once daily for 2 years.

Quality of life is assessed 1 week prior to study drug administration and at 6, 12, 24 and 36 months after study drug administration.

Participants are followed for 1 year.

PROJECTED ACCRUAL: A total of 41 participants will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At risk for developing invasive breast cancer by virtue of 1 of the following criteria:

  * Gail model risk equal to that of an average 60 year old woman as determined using the Gail risk assessment model
  * Lobular neoplasia
  * Atypical ductal hyperplasia with a positive family history of breast cancer
  * Ductal carcinoma in situ previously treated with mastectomy or lumpectomy and radiation
  * BRCA1 or BRCA2 mutation-positive genotyping
  * Family history consistent with hereditary cancer syndrome of increased breast cancer risk defined as 1 of the following:

    * Family with more than 2 breast cancer cases and one or more cases of ovarian cancer diagnosed at any age
    * Family with more than 3 breast cancer cases diagnosed before age 50
    * Sister pairs with 2 breast cancers, 2 ovarian cancers, or 1 breast and 1 ovarian cancer diagnosed before age 50
* Premenopausal

  * Menstrual cycle of 26-35 days
  * No change in menstrual pattern within the past 6 months (no irregularities)
  * FSH level less than 20 mIU/mL
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 23 to 47

Sex

* Female

Menopausal status

* Premenopausal

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* No history of bleeding disorder

Hepatic

* No history of cirrhosis of the liver
* SGOT/SGPT no greater than 3 times upper limit of normal (ULN)

Renal

* Creatinine no greater than 1.7 mg/dL

Cardiovascular

* No history of pulmonary embolism or deep venous thrombosis

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile participants must use effective non-hormonal contraception (e.g. barrier methods, spermicides, or surgical methods) during and for 3 months after study
* No history of infertility with a suspected ovarian etiology or recurrent ovarian cysts
* No allergy to raloxifene
* No dysfunctional uterine bleeding
* No menorrhagia
* No cervical dysplasia or significant uterine pathology requiring concurrent surgery
* No medical or psychiatric disorder that would preclude study participation
* Normal CA 125 levels

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* At least 6 months since prior steroid therapy (e.g., tamoxifen, estrogen, DHEA, anabolic steroids, or oral contraceptives)

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics
* No prior hysterectomy

Ages: 23 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1998-12; Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Eng-Wong, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Medicine Branch, Bethesda, Maryland, United States

REFERENCES:
- [Result] Eng-Wong J, Orzano-Birgani J, Chow CK, Venzon D, Yao J, Galbo CE, Zujewski JA, Prindiville S. Effect of raloxifene on mammographic density and breast magnetic resonance imaging in premenopausal women at increased risk for breast cancer. Cancer Epidemiol Biomarkers Prev. 2008 Jul;17(7):1696-701. doi: 10.1158/1055-9965.EPI-07-2752. Epub 2008 Jun 26. PMID 18583470
- [Result] Orzano JA, Prindiville S, Zujewski J, et al.: Mammographic density is not modulated by raloxifene in pre-menopausal women at high-risk for invasive breast cancer. [Abstract] Breast Cancer Res Treat 88 (Suppl 1): A-4035, 2004.
- [Result] Eng-Wong J, Hursting SD, Venzon D, Perkins SN, Zujewski JA. Effect of raloxifene on insulin-like growth factor-I, insulin-like growth factor binding protein-3, and leptin in premenopausal women at high risk for developing breast cancer. Cancer Epidemiol Biomarkers Prev. 2003 Dec;12(12):1468-73. PMID 14693739
- [Result] Eng-Wong J, Stratton P, Forman M, et al.: Effect of raloxifene on menstrual cycle length and quality of life in premenopausal women at high risk for invasive breast cancer. [Abstract] American Association for Cancer Research: Frontiers in Cancer Prevention Research, October 26 - 30, 2003, Phoenix, AZ. 12: A-193, 1300s, 2003.
- [Result] Premkumar A, Stratton P, Johnson D, et al.: Long term effects of raloxifene on the ovary and uterus in pre-menopausal women at high risk for developing breast cancer. [Abstract] Ultrasound Obstet Gynecol 22 (Suppl 1): A-OC164, 44, 2003.
- [Result] Premkumar A, Stratton P, Avila N, et al.: Raloxifene effects on the ovary and the uterus in premenopausal subjects at high risk for developing breast cancer - sonographic evaluation. [Abstract] Ultrasound Obstet Gynecol 20 (Supp 1): A-P174, 72, 2002.
- [Result] Zujewski J, Eng-Wong J, Reynolds J, et al.: A phase 2 trial of raloxifene in premenopausal women at high risk for developing invasive breast cancer. [Abstract] Breast Cancer Res Treat 76 (Suppl 1): A-417, 2002.